CLINICAL TRIAL: NCT00593281
Title: INcreased Flow Utilizing Subcutaneously Enabled Morphine (INFUSE-Morphine) With and Without Human Recombinant Hyaluronidase (HYLENEX) and Intravenously
Brief Title: INFUSE Morphine Study
Acronym: INFUSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Richard Yocum, M.D., Halozyme Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HZ2-05-06; 05-015-MI (Hospice #)
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Pain
Keywords: Hyaluronidase; Hylenex; subcutaneous; morphine; absorption; bioavailability; PK study of morphine in patients with pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): IV Morphine
- 2 (Experimental): SC Morphine with Hylenex
  Interventions: Drug: Hylenex
- 3 (Active Comparator): SC Morphine with Saline
  Interventions: Drug: Hylenex

INTERVENTIONS:
Drug: Hylenex — Add Hylenex to SC injection of Morphine
  Arms: 2; 3

SUMMARY:
Double-blind study comparing the pharmacokinetics, safety and tolerability of morphine administered subcutaneously (SC) with and without human recombinant hyaluronidase (HYLENEX) and intravenously conducted in patients in a hospice care setting or through a palliative care medicine setting. In this within-patient controlled study, each eligible study patient receives a single injection by each of the three methods of morphine administration, sequentially on three consecutive days, according to the order specified by a randomization schedule.

Each of the three injections consists of 5 mg of morphine (1.0 mL of 5 mg/mL solution). The HYLENEX injection will be 1 mL of 150 units. Although the IV administration will not be blinded, the two SC injections will be double-blinded, using the same volume of normal saline (0.9% sodium chloride) placebo (1.0 mL) as HYLENEX.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females at least 18 years of age who are patients of San Diego Hospice & Palliative Care or recruited through San Diego Hospice & Palliative Care or the UCSD Center for Pain and Palliative Medicine.
2. During the treatment days of the study, on opioid therapy other than morphine that is equivalent to ≥ 60 mg oral morphine per day and without unacceptable toxicity.
3. Vital signs (BP, HR, RR) within normal range.
4. Adequate venous access in both upper extremities.
5. A negative pregnancy test (if female of child-bearing potential) within 7 days prior to first injection.
6. Life expectancy ≥ ten days.
7. Decision-making capacity.
8. Signed, written IRB-approved informed consent. -

Exclusion Criteria:

1. Known hypersensitivity or history of any toxicity to morphine.
2. Morphine within the 4 days prior to the first study medication injection or anticipated to be receiving morphine during any of the treatment days in this study.
3. Any contraindication to morphine.
4. Known hypersensitivity to naloxone.
5. Known allergy to hyaluronidase or any other ingredient in the formulation of HYLENEX.
6. Known allergy to bee or vespid venom.
7. Contraindication to IV heparin lock or known hypersensitivity to heparin.
8. Edema, infection, or any other lower extremity or pelvic disorder that might affect subcutaneous absorption from the thigh.
9. Hemoglobin < 10 g/dL.
10. Presence of any other medical condition that would present an unacceptable safety risk to the patient.
11. Participation in a study of any investigational drug or device within 30 days of enrollment in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
• Determine the Tmax and other pharmacokinetic parameters of morphine injected subcutaneously with HYLENEX compared to without HYLENEX and injected intravenously | 29 days

SECONDARY OUTCOMES:
Compare the safety and tolerability of these three methods of injections of morphine | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Jay Thomas, M.D., Principal Investigator — San Diego Hospice; Mark S Wallace, M.D., Principal Investigator — UCSD Thornton Hospital
Locations (2):
- United States (2):
  - UCSD Thornton Hospital, San Diego, California
  - San Diego Hospice and Palliative Care, San Diego, California

REFERENCES:
- [Derived] Thomas JR, Wallace MS, Yocum RC, Vaughn DE, Haller MF, Flament J. The INFUSE-Morphine study: use of recombinant human hyaluronidase (rHuPH20) to enhance the absorption of subcutaneously administered morphine in patients with advanced illness. J Pain Symptom Manage. 2009 Nov;38(5):663-72. doi: 10.1016/j.jpainsymman.2009.03.009. Epub 2009 Oct 12. PMID 19819665